CLINICAL TRIAL: NCT04372030
Title: Utilisation de Soins Pendant la Crise Covid-19 : Recours, Report et Renoncement (US3R)
Brief Title: Health Care Use During the Covid19 Crisis
Acronym: US3R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: US3R
Record Dates: First submitted 2020-04-22; First posted 2020-05-01 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Health Care Utilization
Keywords: foregone care; postponed care; covid19; confinement
MeSH Terms: conditions — Patient Acceptance of Health Care; COVID-19

STUDY DESIGN:
Intervention Model Description: This is an online survey completed by participants willing to take part
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- General population (Other): There is only one arm wishing to participate
  Interventions: Other: Online questionnaire

INTERVENTIONS:
Other: Online questionnaire — this is an online questionnaire collecting retrospective data on health care use and non-use

SUMMARY:
The project US3R is a general population survey that will measure the magnitude of utilised, postponed and foregone medical care in relation with other health care needs than coronavirus symptoms during the confinement period in Belgium. The study aims to describe the magnitude of unsatisfied health care needs for various types of care. It will also identify the reasons for these postponed and foregone care according to gender, health and socioeconomic status.

DETAILED DESCRIPTION:
Context:

Belgium has put in place confinement measures on March 13th 2020 with the aim to reduce contagion related to Covid19 in the population and manage the number of patients to be treated in the hospital.

However, some weeks after those confinement measures, health care professionals are worry about other patients than Covid19 since they have observed a significantly lower use of emergency services, cancellations of screening appointments, interrupted health care in patients with chronic conditions, disabilities, or mental health disorders.

Objectives: to collect data on used, postponed and foregone medical care related to other health care needs than Covid19 during the confinement period in Belgium; to measure the magnitude of unsatisfied health care needs for various types of care; to identify the reasons explained postponed and foregone care

Methods : the survey is made of about 50 questions collecting self-reported data on health care use and non-use for various types of care along with demographics, socioeconomics and health status characteristics during the confinement period . Data will be analysed with Stata 15 using statistical tests and regression models.

Participants are collected via social media platforms and institutionnal mailing, and Belgian newspapers.

ELIGIBILITY:
Inclusion Criteria:

* living in Belgium
* more than 18

Exclusion Criteria:

* living outside Belgium
* less than 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3164 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Health care use | throughout the whole study, assessed up to 18 months
  Number of person reporting that they used health care during confinement (yes/no)
Postponed heath care use | throughout the whole study, assessed up to 18 months
  Self-reported postponed health care use (yes/no)
Foregone health care use | throughout the whole study, assessed up to 18 months
  Self-reported foregone health care use (yes/no)

CONTACTS AND LOCATIONS:
Locations (1):
- UCLouvain, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No